CLINICAL TRIAL: NCT03312478
Title: To Evaluate the Association Between Type 1 Diabetes Mellitus (T1DM) in Offspring With Positive Parental History of Diabetes
Brief Title: Association of Type 1 Diabetes Mellitus in Offsprings With Positive Parental History of Diabetes
Acronym: SHINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTUL08473; U1111-1200-1995 (Other: UTN)
Record Dates: First submitted 2017-09-29; First posted 2017-10-17 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Case (Other): Known cases of type 1 diabetes mellitus as described in the inclusion criteria for cases
  Interventions: Drug: Blood draw for insulin auto-anti body tests*
- Control (Other): Age-matched non-diabetic controls as described in the inclusion criteria for controls
  Interventions: Drug: Blood draw for insulin auto-anti body tests*

INTERVENTIONS:
Drug: Blood draw for insulin auto-anti body tests* — Pharmaceutical form: N/A
  Route of administration: N/A

SUMMARY:
Primary Objective:

To measure the association between a parental history of diabetes and the odds of an offspring being Type 1 diabetics.

Secondary Objectives:

* To document the profile of Type 1 diabetes patients.
* To document the glycemic parameters (Fasting blood glucose [FBG] and glycosylated hemoglobin [HbA1c]) of Type 1 diabetes.
* To capture the current therapeutic management.

DETAILED DESCRIPTION:
The overall duration of this study is expected to be 12 months. The recruitment period for a given center will be four months following site initiation of that center. telephonic follow-up for all the patients shall be conducted after 15 days ± 5 days.

*Each patient (cases as well as controls) will be required to undergo laboratory tests for insulin autoantibodies and hemoglobin A1c tests. Both the tests will be conducted through centralized laboratories for all recruited patients.

Since the result of insulin auto-antibodies test is one of the inclusion criteria, it is mandatory for all patients to undergo this test, and detailed information for the same has been included in the informed consent form.

ELIGIBILITY:
Inclusion criteria :

Inclusion Criteria for Cases

* Age ≥ 2 years and ≤ 20 years.
* Type 1 diabetes mellitus (T1DM) at any stage of life assessed as:
* Insulin initiated within one year of diagnosis.
* One or more islet autoantibodies (insulin auto-antibodies [IAA], glutamic acid decarboxylase (GAD), or IA2) positive at the time of enrolment. The laboratory value for IAA ≥ 2.4 units/mL, ≥ 10 IU/mL for IA2 and ≥ 5 IU/mL for anti-GAD to be labelled as positive.
* Consenting to participate in the study or care giver ready to sign data release consent if the patient is less than legal limit which is 18 years of age.

Inclusion Criteria for Controls

* Age ≥ 2 years and ≤ 20 years. Every control will be matched for a specific patient within ± two years of age.
* Non diabetic.
* All islet autoantibodies negative at the time of enrolment (IAA, GAD, or IA2). The laboratory value for IAA ≤ 2.4 units/mL, ≤ 10 IU/mL for IA2, and ≤ 5 IU/mL for anti-GAD to be labelled as negative.
* Consenting to participate in the study or care giver ready to sign data release consent if the patient is less than 18 years of age.

Exclusion criteria:

Exclusion Criteria for Cases:

* Age ≤ 2 years and >20 years.
* Patients with any other pre-existing auto-immune disease.
* Gestational Diabetes.
* Pregnant Woman.

Exclusion Criteria for Controls:

* Age ≤ 2 years and > 20 years.
* Patient with history of Type 1 (T1) and Type 2 Diabetes Mellitus (T2DM).
* History of T1 and T2DM in siblings.
* Gestational Diabetes.
* Pregnant Woman.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 375 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2018-08-19 (Actual)

PRIMARY OUTCOMES:
Odds of Type 1 Diabetes Mellitus child having a diabetic parent | 12 months
  Odds ratio will be used to calculate and measure disease frequency from dichotomous categorical variables

SECONDARY OUTCOMES:
Characterization of this population by gender | 12 months
  Categorical variables (gender) will be presented as proportions
Characterization of this population by age | 12 months
  Categorical variables (age) will be presented as proportions
Characterization of this population by socio-economic profile | 12 months
  Categorical variables (socio-economic profile) will be presented as proportions
Means of HbA1c in Type 1 diabetes mellitus (T1DM) patients | 12 months
  Mean HbA1c
Standard deviation of HbA1c in T1DM patients | 12 months
  Standard deviation of HbA1c
Distribution of prescribed therapies by type of insulin to T1DM patients | 12 months
  Distribution of prescribed therapies by type of insulin will be presented as proportions
Means of fasting blood glucose (FBG) in T1DM patients | 12 months
  Mean Fasting Blood Glucose
Standard deviation of FBG in T1DM patients | 12 months
  Standard deviation of FBG
Duration of diabetes in parent | 12 months
  Mean duration of diabetes in parent
Mean duration of diabetes in parent | 12 months
  Standard deviation of duration of diabetes in parent
Characterization of family history of diabetes | 12 months
  Categorical variables will be measured as proportions
Characterization of frequency of consultation | 12 months
  Number of consultations per month
Characterization of diabetes education | 12 months
  Number of sessions per month

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- National Institute of Child Health, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org